CLINICAL TRIAL: NCT01370148
Title: A Phase 1, Open-Label Study to Assess the Effect of Severe Hepatic Impairment on the Pharmacokinetics of Intravenous Conivaptan
Brief Title: A Study to Assess the Effect of Severe Hepatic Impairment on the Pharmacokinetics of Intravenous Conivaptan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 087-CL-099
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Liver Disease
Keywords: Pharmacokinetics; Protein Binding; Conivaptan; Vaprisol; Liver Disease; YM087
MeSH Terms: conditions — Liver Diseases | interventions — conivaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects with severe hepatic impairment (Experimental)
  Interventions: Drug: conivaptan hydrochloride
- Subjects with normal hepatic function (Active Comparator)
  Interventions: Drug: conivaptan hydrochloride

INTERVENTIONS:
Drug: conivaptan hydrochloride — Intravenous
  Other Names: Vaprisol; YM087

SUMMARY:
The purpose of this study is to assess the pharmacokinetics and safety of a 48-hour continuous infusion of conivaptan in subjects with severe liver impairment compared to subjects with normal liver function.

DETAILED DESCRIPTION:
Subjects will be admitted to the Phase 1 unit Day -2 and will remain confined to the unit until discharge on Study Day 5 after completion of all study procedures.

ELIGIBILITY:
Inclusion Criteria:

Subjects with Normal Hepatic Function:

Female subject must be either:

* post-menopausal prior to Screening, or
* premenarchal prior to Screening, or
* documented surgically sterile or post hysterectomy, or
* if of childbearing potential, must have a negative pregnancy test at Screening and must be using highly effective contraception prior to Screening and throughout the study period and for 28 days after final study drug administration

  * Female subject must not be lactating and must not be breastfeeding at Screening or during the study period, and for 28 days after final study drug administration
  * Female subject must not donate ova starting at Screening or during the study period, and for 28 days after final study drug administration
  * Male subject must:
* be using highly effective contraception consisting of two forms of birth control (one of which must be a barrier method) starting at Screening and continue throughout the study period, and for 28 days after final study drug administration
* not donate sperm starting at Screening and throughout the study period, and for at least 28 days after final study drug administration

  * Subject weighs at least 45 kg and has a body mass index between 18 and 40 kg/m2 inclusive
  * The subject must have clinical laboratory test results within normal range, including liver function tests (LFTs)
  * The subject must have had a normal 12-lead electrocardiogram (ECG)

Hepatic Impaired Subjects:

* Female subject must be either:

  * post-menopausal prior to Screening, or
  * premenarchal prior to Screening, or
  * documented surgically sterile or post hysterectomy, or
  * if of childbearing potential, must have a negative pregnancy test at Screening and must be using highly effective contraception prior to Screening and throughout the study period and for 28 days after final study drug administration
* Female subject must not be lactating and must not be breastfeeding at Screening or during the study period, and for 28 days after final study drug administration
* Female subject must not donate ova starting at Screening or during the study period, and for 28 days after final study drug administration
* Male subject must:

  * be using highly effective contraception consisting of two forms of birth control (one of which must be a barrier method) starting at Screening and continue throughout the study period, and for 28 days after final study drug administration
  * not donate sperm starting at Screening and throughout the study period, and for at least 28 days after final study drug administration
* Subject meets criteria for severe hepatic impairment defined by Child-Pugh method
* Subject weighs at least 45 kg and has a body mass index between 18 and 40 kg/m2 inclusive
* The subject must have clinical laboratory test results within therapeutic range except for hepatic disease
* The subject must have had a normal 12-lead electrocardiogram (ECG)

Exclusion Criteria:

Subjects with Normal Hepatic Function:

* Subject has a history of a clinically significant illness, and associated clinical symptoms, medical condition, or laboratory abnormality within past 3 months that would preclude participation in the study
* Subject has evidence of biliary obstruction or other causes of hepatic impairment
* Subject is known to have hepatitis or is a carrier of hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or is known to be HIV positive or has HIV antibodies
* Subject has an impaired ability to sense thirst
* Subject has serum sodium less than 115mEg/L or greater than 140 mEg/L
* Subject has either a systolic blood pressure (BP) of greater than 140 mmHg or a diastolic BP of less than 56 mmHg
* Subject has taken any prescription or over-the-counter medications except for contraceptives, hormone replacement therapy and occasional acetaminophen, or alternative and complementary medicines within past 14 days
* Subject has a history of carcinoma, except for basal cell or cutaneous squamous cell carcinoma within past 5 years
* Subject drinks greater than 14 units of alcohol per week (Note: one unit = 12 ounces of beer, 4 ounces of wine, or 1 ounce of spirits)
* Subject has a history of substance abuse within past 6 months prior to Screening Visit or the subject tests positive at Screening or clinic admission for alcohol or drugs of abuse
* Subject is currently participating in another clinical trial or has received an investigational medication within past 30 days
* Subject is known to have hypersensitivity to conivaptan or its derivatives
* Subject has had a blood transfusion or donated/lost more than 550ml of blood within past 8 weeks
* Subject is incapable of being compliant with the protocol

Subjects with Hepatic Impairment:

* Subject has a history of a clinically significant illness, and associated clinical symptoms, medical condition, or laboratory abnormality within past 3 months that would preclude participation in the study. Subjects with controlled hypertension may be allowed
* Subject has a condition associated with hepatic disease including; biliary obstruction, or other cause of hepatic impairment not related to parenchymal disorder and/or disease of the liver, fluctuating or rapidly deteriorating hepatic function, biliary liver cirrhosis, history or presence of hepatic encephalopathy greater than Grade 1 within past 3 months or unstable encephalopathy prior to Screening, tense ascites, esophageal/gastric variceal bleeding with past 6 months, server portal hypertension, surgical portal systemic shunt or peritoneal venous shunt, thrombocyte level below 50,000 x 10^9/L and prothrombin time (PT) above 18 seconds
* Subject is hypovolemic or has evidence of orthostatic hypotension
* Subject has an impaired ability to sense thirst
* Subject has serum sodium less than 115mEg/L or greater than 140 mEg/L
* Subject has either a systolic blood pressure (BP) of greater than 140 mmHg or a diastolic BP of less than 56 mmHg
* Subject is known to be HIV positive or has HIV antibodies
* Subject has had a change in dose regimen of medication needed for their underlying medical condition with the past four weeks
* Subject is currently taking a prohibited medication
* Subject drinks greater than 14 units of alcohol per week (Note: one unit equals 12 ounces of beer, 4 ounces of wine, or 1 ounce of spirits)
* Subject has a history of substance abuse within past 6 months prior to Screening Visit or the subject tests positive at Screening or clinic admission for alcohol or drugs of abuse
* Subject is currently participating in another clinical trial or has received an investigational medication with past 30 days
* Subject has had a blood transfusion or donated/lost more than 550ml of blood within past 8 weeks
* Subject is known to have hypersensitivity of conivaptan or its derivatives
* Subject is incapable of being compliant with the protocol

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Assess the effect of severe hepatic impairment on the plasma drug concentration of conivaptan through analysis of blood samples | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Art Wheeler, MD, Study Director — Cumberland Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Advanced Clinical Research Institute, Anaheim, California
  - DaVita Clinical Research, Lakewood, Colorado
  - Orlando Clinical Research, Orlando, Florida